CLINICAL TRIAL: NCT05247281
Title: Randomized Controlled Trial Investigating the Use of Next-generation Sequencing in Directing the Antimicrobial Treatment of Periprosthetic Joint Infection
Brief Title: NGS vs Culture Outcomes for Treatment of PJI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Center for Innovation and Research Organization (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022NGSOutcomes
Record Dates: First submitted 2022-01-13; First posted 2022-02-18 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-10

CONDITIONS: Prosthetic Joint Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Culture-based treatment (Active Comparator)
  Interventions: Diagnostic Test: Culture-based treatment
- Next Generation Sequencing (NGS) with Culture-based treatment (Active Comparator)
  Interventions: Diagnostic Test: Next Generation Sequencing (NGS) with Culture

INTERVENTIONS:
Diagnostic Test: Culture-based treatment — Medications to treat prosthetic joint infection will be chosen based on results of traditional cultures alone
  Arms: Culture-based treatment
Diagnostic Test: Next Generation Sequencing (NGS) with Culture — Medications to treat prosthetic joint infection will be chosen based results of NGS and culture
  Arms: Next Generation Sequencing (NGS) with Culture-based treatment

SUMMARY:
This multicenter, randomized controlled trial will compare the use of NGS and traditional culture in directing antimicrobial treatment for patients with periprosthetic joint infection.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age > 18 years)
* Undergoing single stage revision or 1st stage resection arthroplasty/spacer placement for PJI (ICM-positive) of the hip or knee
* Written informed consent

Exclusion Criteria:

* Ongoing participation in another clinical trial
* Megaprosthesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants who have been diagnosed with prosthetic joint infection as assessed by the 2018 International Consensus Definition of prosthetic joint infection | 90 days from time of surgery
  Diagnosis of re-infection following surgery and treatment for prosthetic joint infection

SECONDARY OUTCOMES:
Number of subjects who have a re-operation as assessed by inpatient hospitalization medical records | one year from time to surgery

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Morrison, Study Director — Center for Innovation and Research Organization
Locations (9):
- United States (9):
  - University of Southern California, Los Angeles, California
  - Cleveland Clinic Florida, Weston, Florida
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University, New York, New York
  - University of Rochester, Rochester, New York
  - Northwell Health, Staten Island, New York
  - Cleveland Clinic Ohio, Cleveland, Ohio
  - Rothman Orthopaedic Institute, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah